CLINICAL TRIAL: NCT00065936
Title: Behavioral and Biochemical Mechanisms of Self-Injury
Brief Title: Self-Injury: Diagnosis and Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R29HD35862; R29 HD35862; NICHD-0525
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Self-Injurious Behavior; Mental Retardation
Keywords: Intractable self-injurious behavior; Naltrexone; Transcutaneous electrical nerve stimulation; Substance P; Met-enkephalin; Cortisol
MeSH Terms: conditions — Self-Injurious Behavior; Intellectual Disability | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone hydrochloride
Procedure: Transcutaneous sensory nerve stimulation

SUMMARY:
Self-injurious behavior is behavior in which a person hurts or harms himself. This behavior sometimes occurs in people with mental retardation or autism. This study will evaluate self-injurious behavior in people with mental retardation or autism and will test the effectiveness of new treatments.

DETAILED DESCRIPTION:
It is unknown why some people with mental retardation and/or autism repeatedly and persistently injure themselves, some to the point of tissue damage and permanent scarring. Unraveling this mystery poses paradoxical biomedical and behavioral science questions and creates deeply troubling problems for practitioners and family members of affected individuals. Over the past decade, many cases of self-injurious behavior (SIB) have been treated successfully using behavioral interventions that teach communication and other functional skills. However, practical problems of implementation, costs associated with long-term treatment, and cases with no clear social profile suggest that there is still much to be learned about why people self-injure. Some forms of self-injury may involve intense stimulation of body sites sufficient to elicit the release and receptor binding of endogenous opioid peptides. This study will evaluate variables common to SIB and the neurophysiology of pain regulation. The study will also clarify the role of the endogenous opioids and pain mechanisms in self-injury.

Participants with mild to profound mental retardation and/or autism will be observed for frequency of self-injury, duration and intensity of self-injurious behavior, and where on the body that behavior is directed. Following this characterization, participants' saliva will be noninvasively examined for substance P, met-enkephalin, and cortisol as markers for altered pain transmission and predictors of response to treatment. After screening and SIB subtyping (i.e., social, nonsocial, or mixed), 37 participants whose self-injury is primarily nonsocial or mixed will be evaluated over 16 weeks. Participants will be randomized to receive either transcutaneous electric nerve stimulation (TENS, an opioid agonist treatment) or naltrexone (an opioid antagonist treatment). Participants whose self-injury is primarily socially motivated will be evaluated with TENS and will receive behavioral interventions through a technical assistance service delivery model. Follow-up evaluations will occur at Months 3 and 6.

ELIGIBILITY:
Inclusion Criteria

* Self-injurious behavior for at least 3 months prior to study entry
* Normal cardiac, liver, and kidney function as determined by a physician

Exclusion Criteria

* Only presenting problems are pica, aggression, property destruction, hyperkinesis, screaming, or eating disorders
* Lesch-Nyhan syndrome
* Peripheral neuropathy
* Self-injury that presents immediate imminent risk such as loss of sight or hearing or other potentially life threatening behavior
* Serious chronic health impairments associated with specific syndromes (e.g., Cornelia de Lange, Prader Willi Syndrome)
* Self-injury unresponsive to prior conventional behavioral or pharmacological interventions (e.g., less than 50% reduction in overall self-injury for 3 months)
* Major depressive disorder or schizophrenia

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37
Dates: Start 1997-07; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Frank Symons, Ph.D., Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - Frank Porter Graham Child Development Center, University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Research Training Institute, Western Carolina Center, Morganton, North Carolina

REFERENCES:
- [Background] Symons FJ, Koppekin A, Wehby JH. Treatment of self-injurious behavior and quality of life for persons with mental retardation. Ment Retard. 1999 Aug;37(4):297-307. doi: 10.1352/0047-6765(1999)0372.0.CO;2. PMID 10463024
- [Background] Symons FJ, Sutton KA, Walker C, Bodfish JW. Altered diurnal pattern of salivary substance P in adults with developmental disabilities and chronic self-injury. Am J Ment Retard. 2003 Jan;108(1):13-8. doi: 10.1352/0895-8017(2003)1082.0.CO;2. PMID 12475363
- [Background] Breau LM, Camfield CS, Symons FJ, Bodfish JW, Mackay A, Finley GA, McGrath PJ. Relation between pain and self-injurious behavior in nonverbal children with severe cognitive impairments. J Pediatr. 2003 May;142(5):498-503. doi: 10.1067/mpd.2003.163. PMID 12756380